CLINICAL TRIAL: NCT01373827
Title: Protocol To Evaluate Patient Measurements After Ultrasonic Treatment.
Status: Completed | Type: Observational
Sponsor: Sound Surgical Technologies, LLC. (Industry)
Responsible Party: Roy G Geronemus, MD, Laser & Skin Surgery Center of New York
Other Study IDs: SST2011-2
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Patients Treated With VaserShape MC1
Keywords: VASER; VASERShape; MC1; ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MC1 Subjects
  Interventions: Device: VASERShape MC1

INTERVENTIONS:
Device: VASERShape MC1 — Use of the VASERShape MC1 device as part of routine practice

SUMMARY:
Patients enrolled in this study will come from the Investigator's patient population and be ordinarily suitable for treatment using the MC1 device. The treatment they receive will be no different if they participate than if they do not. The study is only to observe the patients before, during and after their usual treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Female between 20 and 50 years of age, inclusive, on the day of enrolment.
2. Has a BMI between 20 and 30 kg/m2.
3. Is to be treated in the posterior thigh / saddlebag area using the MC1.
4. Has never been treated with the MC1 before.
5. Females who are post menopausal or using a medically acceptable form of birth control prior to study enrollment and during the course of the study. (i.e., condoms with spermicide, oral contraceptives contraceptive implants etc.)

Exclusion Criteria:

1. Subject is lactating, has a positive pregnancy test within 7 days of planned study procedure (for female subjects of child-bearing potential), or intends to become pregnant during the study.
2. Currently enrolled in another device or drug study that has not completed the required follow-up period, or has completed all other study-required follow-up less than 30 days before enrolment in this study.
3. Keloid scars, hypertorphic scars or a history of abnormal healing.
4. Any known bruising disorder, anticoagulative / thromboembolic condition , hemorrhagic (bleeding) status or use of anti coagulants.
5. Tissue ischemia in the area to be treated.
6. Suffering from concurrent conditions such as liver or kidney disorders, Hypertension or abnormally high blood pressure.
7. High cholesterol and/or diabetes.
8. Active collagen vascular disease (e.g. fibromyalgia, panniculitis, lupus etc.).
9. Epilepsy.
10. Tuberculosis.
11. Auxiliary electric organs (such as pacemakers), metal or myoelectric prosthesis.
12. Suffering from Endocrine syndromes or thyroid hyperfunction.
13. Active skin infection, any infection in the treated area within the last 30 days or skin disease in the area to be treated (e.g. eczema, psoriasis, urticaria, dermographism).
14. Bone, muscle or joint disease, dysfunction or healing in the area to be treated.
15. Malignancy in the area to be treated.
16. Laminectomy in the area to be treated.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All subjects presenting to the investigator for treatment using the MC1 are potential study candidates and will be screened for eligibility. Every effort will be made to establish eligibility of the participants before enrollment. Subjects who do not meet all inclusion/exclusion criteria will not be enrolled. Enrollment in the study occurs at the time the patient is randomized to the assigned treatment.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laser & Skin Surgery Center of New York, New York, New York, United States